CLINICAL TRIAL: NCT06117930
Title: Study of Human Brain-Gut Axis and Gut Microbiome In Patients With Brain Lesions - Repository for Neuroscience Research
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC230707; NCI-2023-04797 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-001388 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Malignant Central Nervous System Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples stored for future research if participant gives permission.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Participants undergo blood, tissue, saliva, urine and stool sample collection and complete questionnaires on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study explores how microorganisms in the gut can affect the growth and progression of brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish a Mayo Clinic Florida Brain Tumor-Gut Axis Human Biorepository by sequential collection of fecal, urine, blood, saliva, and/or tissue samples and clinical patient information.

II. To use spatial transcriptome/proteomics/multi-omics coupled with microbiome data from various sources including brain tissue and stool samples to understand how microbiota could impact disease development, progression, and treatment response in patients with brain cancer.

III. To study the effect of microbiome and potential relationships and/or microbiome reconstruction to impact patient's clinical outcomes including chemo, radiation, immunotherapy and/or cellular therapy.

OUTLINE: This is an observational study.

Participants undergo blood, tissue, saliva, urine and stool sample collection and complete questionnaires on study.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing resection for a tumor of the central nervous system and associated controls are eligible to participate in this study.

Exclusion Criteria:

* Excluded samples will be from patients younger than 18 years old. There are no exclusions due to race/sex.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing resection for a tumor of the central nervous system and associated controls are eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2029-12-13 (Estimated); Study Completion 2029-12-13 (Estimated)

PRIMARY OUTCOMES:
Establish the Mayo Clinic Florida Tumor-Gut Axis Biorepository | Approximately 1 year, or until samples have been collected based on scheduled treatment.
  Biological samples such as stool, urine, blood, saliva, and/or tissue will be collected for storage in the Tumor-Gut Axis Biorepository. Samples may be collected at any of the following time periods during study participation: before/after steroid therapy, before/after surgical intervention, before/after radiation therapy, and before/after chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Quinones-Hinojosa, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials